CLINICAL TRIAL: NCT01888289
Title: An Open Label, Randomized, Single Dose, Oral Bioequivalence Study of Isotretinoin Capsules 40 mg of Dr. Reddy's Laboratories Limited, India Comparing With That of ACCUTANE® Capsules 40 mg of Roche Laboratories Inc., Under Fasting Conditions
Brief Title: Bioequivalence Study of Isotretinoin Capsules 40 mg Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AAI-US-101
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2001-11

CONDITIONS: Healthy
MeSH Terms: interventions — Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isotretinoin capsules, 40 mg (Experimental): Isotretinoin Capsules, 40 mg of Dr.Reddy's Laboratories Ltd
  Interventions: Drug: Isotretinoin
- ACCUTANE (Active Comparator): ACCUTANE 40 mg of Roche Laboratories Inc
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Drug: Isotretinoin — Isotretinoin Capsules,40 mg
  Other Names: ACCUTANE

SUMMARY:
The purpose of this study is to determine the pharmacokinetics and bioequivalence of isotretinoin formulations after administration of single doses to normal, non-smoking,healthy males under fasting conditions

DETAILED DESCRIPTION:
An open label, randomized, two-treatment, single dose, oral bioequivalence study of Isotretinoin capsules 40 mg of Dr. Reddy's Laboratories Limited,under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males between 18 and 45 years of age inclusive.
2. Informed of the nature of the study and given written informed consent.
3. Have a body weight within 15% of the appropriate range as defined in the 1983 Metropolitan Life Company tables and weighing at least 125 lbs. (Appendix I).

Exclusion Criteria

1. Hypersensitivity to isotretinoin or related compounds.
2. Any history of a clinical condition which might affect drug absorption, metabolism or excretion.
3. Recent history of mental illness, drug addiction, drug abuse or alcoholism.
4. Donation of greater than 500 ml of blood in the past 4 weeks prior to study dosing or difficulty in donating blood.
5. Received an investigational drug within the 4 weeks prior to study dosing.
6. Currently taking any prescription medication within the 7 days prior to study dosing or over-the-counter medication within 3 days of study dosing. This prohibition does not include vitamins or herbal preparations taken as nutritional supplements for non-therapeutic indications as judged by the attending physician.
7. Regular tobacco use in the 3 months prior to study dosing.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2001-07; Primary Completion 2001-08 (Actual); Study Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) | Pre-dose (0) and 0.5, 1,2,3,4,5,6,8,10,16,24,36,48,72 and 96hrs

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ralph Scallion, MD, Principal Investigator — AAI
Locations (1):
- AAI, Quadrangle Drive, Chapel Hill,, North Carolina, United States